CLINICAL TRIAL: NCT01708239
Title: Sequential Use of the LEFt Rule, D-dimer Measurement and Complete Ultrasonography to Rule Out Deep Vein Thrombosis During Pregnancy: a Prospective Outcome Study.
Brief Title: Left Rule, D-Dimer Measurement and Complete Ultrasonography to Rule Out Deep Vein Thrombosis During Pregnancy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marc Righini (Other)
Collaborators: University Hospital, Brest (Other); The Ottawa Hospital (Other)
Responsible Party: Sponsor-Investigator, Marc Righini, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: Geneva University Hospital
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy; Deep Vein Thrombosis
Keywords: Pregnancy; Deep vein thrombosis; Clinical probability; D-Dimer; Compression ultrasonography
MeSH Terms: conditions — Venous Thrombosis | interventions — fibrin fragment D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women with suspected DVT assessed by the LEFt rule, D-dimer measurement and complete ultrasonography.
  Interventions: Other: Left rule, D-dimer measurement and complete ultrasonography in pregnant women.

INTERVENTIONS:
Other: Left rule, D-dimer measurement and complete ultrasonography in pregnant women. — Diagnostic strategy based on the LEFt rule, D-dimer measurement and complete ultrasonography

SUMMARY:
In pregnant women with suspected DVT, a sure diagnosis is mandatory. In non-pregnant patients, sequential diagnostic strategies based on 1) the assessment of clinical probability, 2) D-dimer measurement and 3) compression ultrasonography (CUS) have been well validated.

Clinical probability assessment by clinical prediction rules (CPRs) is a crucial step in the management of suspected DVT. However, the most commonly used CPR for DVT, the Wells' score, has never been validated in pregnant women. Recently, the 'LEFt' clinical prediction rule was derived and internally validated. A prospective validation of this rule is now warranted, and we plan to use it in our prospective study.

The second step used in the diagnostic strategy including non-pregnant patients is D-dimer measurement. The test has been widely validated in non-pregnant patients and, in association with a non-high clinical probability, it allows to safely rule out DVT.

As D-dimer level raise steadily during pregnancy, the specificity of the test decreases and it is less useful in pregnant women. Data from the literature clearly suggest that the usual cut-off set a 500 ng/ml would safely rule out DVT in pregnant women [6]. As the usual cut-off has never been prospectively validated in pregnant women with suspected DVT, we would like to use it in our study.

Some studies suggested that complete CUS is safe to rule out DVT in pregnant women. However, this test is not always available. Therefore, a strategy in which the association of clinical probability assessment and D-dimer measurement would allow to safely rule out DVT in a significant proportion of patients without performing a complete CUS, would be of great help in everyday clinical practice and would probably be cost-effective.

Therefore, we plan a prospective study to assess the safety of a sequential diagnostic strategy based on the assessment of clinical probability with the LEFt rule, D-dimer measurement and complete CUS in pregnant women with suspected DVT.

DETAILED DESCRIPTION:
In pregnant women with suspected DVT, a sure diagnosis is mandatory. Indeed, false positive tests lead to inappropriate anticoagulant treatment, which increases the risk of bleeding. Conversely, false negative tests might lead to a life-threatening thromboembolic event. Thus, accuracy of diagnostic methods used in pregnant women is crucial [1].

In non-pregnant patients, sequential diagnostic strategies based on 1) the assessment of clinical probability, 2) D-dimer measurement and 3) compression ultrasonography (CUS) have been widely validated [2, 3].

Clinical probability assessment by clinical prediction rules (CPRs) is a crucial step in the management of suspected DVT. However, the most commonly used CPR for DVT, the Wells' score, has never been validated in pregnant women [3]. Recently, the 'LEFt' clinical prediction rule was derived and internally validated by Chan et al. among 194 pregnant women investigated for suspected DVT[4]. This rule combines three variables: symptoms in the left leg ("L"), calf circumference difference equal or greater than 2 centimeters ("E" for edema) and first trimester presentation ("Ft") [4].

We performed an external validation of this rule on a recently published prospective cohort of pregnant patients with suspected DVT (submitted to JTH). This external validation showed that a negative "LEFt" rule accurately identified pregnant women in whom the proportion of confirmed DVT appears to be very low. A prospective validation of this rule is now warranted, and we plan to use it in our prospective study.

The second step used in the diagnostic strategy including non-pregnant patients is D-dimer measurement. The test has been widely validated in non-pregnant patients and, in association with a non-high clinical probability, it allows to safely rule out DVT [5].

As D-dimer level raise steadily during pregnancy, the specificity of the test decreases and it is less useful in pregnant women. A recent study suggested that the currently available sensitive D-dimer assays that are used for the exclusion in symptomatic non-pregnant women have the potential to exclude DVT in symptomatic pregnant women with the application of higher cut-points [6]. Even if this data arises from a small study, it clearly suggests that the usual cut-off set a 500 ng/ml would safely rule out DVT in pregnant women [6]. As the usual cut-off has never been prospectively validated in pregnant women with suspected DVT, we would like, as a first step, to use it in our study.

In pregnant patients, limited data is available on the use of complete compression ultrasonography to rule out DVT. In a recent prospective management study, we included 226 pregnant and post-partum women with suspected lower limb DVT. We observed a 1.1% (95% CI:0.3-4.0) three-month thromboembolic event rate in those left untreated on the basis of a negative single complete CUS [7]. This result is in line with what was reported after a normal phlebography, the gold standard test [8].

Even if complete CUS is safe to rule out DVT in pregnant women, current diagnostic strategies for suspected DVT in non-pregnant patients rely on the use of clinical probability and D-Dimer prior to leg veins imaging [5]. However, no management outcome study on the safety and usefulness of D-Dimer to rule out DVT in pregnant women is available to date. Another limitation of the strategies based on a single unique complete CUS, is that every woman has to undergo complete CUS. However, this test is not always available. Therefore, a strategy in which the association of clinical probability assessment and D-dimer measurement would allow to safely rule out DVT in a significant proportion of patients without performing a complete CUS, would be of great help in everyday clinical practice and would probably be cost-effective.

Therefore, we plan a prospective study to assess the safety of a sequential diagnostic strategy based on the assessment of clinical probability with the LEFt rule, D-dimer measurement and complete CUS in pregnant women with suspected DVT.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with clinically suspected DVT

Exclusion Criteria:

* Age less than 18
* No available informed consent
* Associated suspicion of pulmonary embolism
* Ongoing anticoagulant treatment
* Planned anticoagulant treatment at therapeutic dosage during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with suspected DVT
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The main outcome will be the number of thromboembolic recurrent events (DVT, PE, death attributable to venous thromboembolic disease) documented during the three-month follow-up in the patients left untreated on the basis of a normal diagnostic strategy. | 3 years
  Rate of thromboembolic events after a normal diagnostic strategy.

SECONDARY OUTCOMES:
Prospective evaluation of the diagnostic performances of the LEFt rule. | 3 years
  Prospective validation of the LEFt rule.
Prospective evaluation of D-dimer measurement to rule out DVT in pregnant women. | 3 years
  Prospective evaluation of the diagnostic performances of D-dimer measurement in pregnant women with suspected DVT.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Le Gal, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- Geneva University Hospital, Geneva, Switzerland